CLINICAL TRIAL: NCT05386784
Title: Effect of Raloxifene Plus Cholecalciferol and Cholecalciferol Alone on the Bone Mineral Density in Postmenopausal Women With Osteopenia: an 1-year Randomized Controlled Trial
Brief Title: Effect of Raloxifene Plus Cholecalciferol and Cholecalciferol Alone on the Bone Mineral Density in Postmenopausal Women With Osteopenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-0977
Record Dates: First submitted 2022-05-18; First posted 2022-05-23 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Postemenopusal Women With Osteopenia
MeSH Terms: interventions — Raloxifene Hydrochloride; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raloxifen plus cholecalciferol (Active Comparator): Raloxifene 60mg + Cholecalciferol 800 IU
  Interventions: Drug: Raloxifene plus cholecalciferol
- Cholecalciferol (Active Comparator): Cholecalciferol 800 IU
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Raloxifene plus cholecalciferol — Rabone D ( Raloxifene 60mg + Cholecalciferol 800 IU ) 1 Capsule once daily
  Other Names: Rabone D
  Arms: Raloxifen plus cholecalciferol
Drug: Cholecalciferol — D3 oral base drop, 4 drops once daily (800 IU)
  Other Names: D3 base oral drop
  Arms: Cholecalciferol

SUMMARY:
Osteoporosis is a very strong predictor of fractures with low BMD, but more than half of osteoporotic fractures actually occur in the osteopenic patient group. Therefore, it is important to prevent fractures by actively evaluating fracture risk even in patients with osteopenia.

Raloxifene is a second-generation SERM agent that inhibits bone resorption and is used for the prevention and treatment of postmenopausal osteoporosis. The clinical effect of raloxifene has already been demonstrated in the Multiple Outcomes of Raloxifene Evaluation (MORE) study, a large-scale RCT, to increase BMD and improve lipid profile. In this study, we aimed to evaluate the efficacy of Raloxifene plus cholecalciferol in postmenopausal women with osteopenia.

DETAILED DESCRIPTION:
Backgroud : Osteoporosis is a powerful predictor of fractures with low BMD, but more than half of osteoporotic fractures occur in osteopenia. Therefore, it is important to start drug treatment after diagnosis of osteoporosis, but it is also important to prevent fractures by actively evaluating the risk of fractures in patients with osteopenia. Raloxifene is a selective oestrogen receptor modulator (SERM) that has beneficial effects on bone and lipid profile and has been approved by the FDA as a treatment to prevent osteoporosis. However, studies on the efficacy of Raloxifene plus cholecalciferol in osteopenia patients lack evidence.

Aim : This study aimed to investigate the efficacy of raloxifene plus cholecalciferol in postmenopausal women with osteopenia.

Methods : A prospective, single-center, randomized, opne label, parallel, intervention study in 112 patients investigating the difference in bone mineral density between raloxifene plus cholecalciferol group and cholecalciferol group. Study participants are randomly assigned using the R procedure in a 1:1 ratio at enrollment. Each participant takes raloxifene plus cholecalciferol or cholecalciferol for 48 weeks. All participants were tested for bone turnover markers, routine chemistry, and lipid profile at baseline and 6-month intervals. In addition, at baseline and 48 weeks, DXA, whole spine x-ray, quantitative CT, bioimpedance analysis, muscle function test (handgrip test, jump power), and EQ-5D test.

Perspectives : More than half of osteoporotic fractures occur in patients with osteopenia. This study will confirm the effect of Raloxifene plus cholecalciferol on bone density and show changes in muscle function and lipid metabolism. Through this, early and active treatment can be suggested as a new guideline for preventing osteoporosis and osteoporotic fractures in postmenopausal women with osteopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women (defined as no menstruation for more than 48 weeks prior to screening and no other pathological or physiological causes. If in doubt, a serum follicle-stimulating hormone (FSH) test may be performed at screening)
2. Osteopenia ( -2.5 SD< T-score < -1.0 SD in DXA )

Exclusion Criteria:

1. Secondary osteoporosis (Systemic glucocorticoid use, aromatase inhibitor, thyrotoxicosis, hypeparathyroidism, etc)
2. Vitamin D deficiency at baseline (25-OH-vitD <10ng/mL)
3. Active cancer treatment
4. History of vascular thrombosis
5. Bisphosphonate treatment within the last 12months
6. Contraindication for Raloxifene according to the SPC

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 112 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
BMD lumbar spine | 48 weeks
  Change in lumbar spine BMD from baseline to 48 weeks after the Ralxifene plus cholecalciferol vs cholecalciferol

SECONDARY OUTCOMES:
BMD femoral neck and total hip | 48 weeks
  Change in femoral neck and total hip BMD from baseline to 48 weeks after the Ralxifene plus cholecalciferol vs cholecalciferol
Bone turnover marker | 24 weeks, 48 weeks
  Changes in p-CTX and P1NP From Baseline to 24 and 48 weeks after the Ralxifene plus cholecalciferol vs cholecalciferol
Muscle function | 24 weeks, 48 weeks
  Changes in muscle fucntion (Handgrip, jump power) From Baseline to 24 and 48 weeks after the Ralxifene plus cholecalciferol vs cholecalciferol
Lipid profile | 24 weeks, 48 weeks
  Changes in lipid profile From Baseline to 24 and 48 weeks after the Ralxifene plus cholecalciferol
Vertebral fracture | 48 weeks
  Morphometric Vertebral Fractures Assessed by whole spine x-ray
Quantitative CT | 48 weeks
  Change in quantitative CT from baseline to 48 weeks after the Ralxifene plus cholecalciferol vs cholecalciferol Morphometric Vertebral Fractures Assessed by whole spine x-ray Baseline to 48 weeks after the Ralxifene plus cholecalciferol vs cholecalciferol
Bioimpedance analysis | 24 weeks, 48 weeks
  Changes in bioimpedance analysis From Baseline to 24 and 48 weeks after the Ralxifene plus cholecalciferol vs cholecalciferol
EQ-5D test | 24 weeks, 48 weeks
  Changes in EQ-5D test From Baseline to 24 and 48 weeks after the Ralxifene plus cholecalciferol vs cholecalciferol

CONTACTS AND LOCATIONS:
Overall Officials: Yumie Rhee, Principal Investigator — Department of Internal Medicine, Endocrine Research Institute, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shin S, Hong N, Rhee Y. A randomized controlled trial of the effect of raloxifene plus cholecalciferol versus cholecalciferol alone on bone mineral density in postmenopausal women with osteopenia. JBMR Plus. 2024 May 30;8(7):ziae073. doi: 10.1093/jbmrpl/ziae073. eCollection 2024 Jul. PMID 38939828